CLINICAL TRIAL: NCT02230410
Title: CryoBalloon Focal Ablation System for Residual Barretts Esophagus Post Ablation; a Pilot Study.
Brief Title: Cryo Balloon for Residual Barrett's Esophagus
Acronym: Cryoballoon
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Pentax Medical (Industry)
Responsible Party: Principal Investigator, Kenneth K. Wang, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-004771
Record Dates: First submitted 2014-08-27; First posted 2014-09-03 (Estimated); Results first posted 2022-02-10 (Actual); Last update posted 2022-02-10 (Actual); Status verified 2022-01

CONDITIONS: Barrett's Esophagus
Keywords: Barrett's; high grade dysplasia; ablation; cyrotherapy
MeSH Terms: conditions — Barrett Esophagus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- focal cryo ablation (Experimental): Subjects with residual barrett's esophagus (less than 3 cm) post ablation will under go one CryoBalloon Focal Ablation treatment
  Interventions: Device: CryoBalloon Focal Ablation

INTERVENTIONS:
Device: CryoBalloon Focal Ablation

SUMMARY:
This study is being done to see if treating residual Barrett's Esophagus after previously having undergone Radiofrequency ablation or Endoscopic Mucosal resection can be eliminated with focal cryotherapy.

ELIGIBILITY:
Inclusion criteria:

* Age > 18 years old
* Able to provide informed consent
* Patients with unifocal or multifocal BE with 2 cm who have failed at least 2 serial RFA or other endoscopic therapy such as Endoscopic Mucosal resection,

Exclusion criteria:

* Age younger than 18 years old
* Presence of esophageal varices
* Esophageal stricture precluding passage of an endoscope
* Inability to provide informed consent
* Esophageal cancer (T2 and above)
* Coagulopathy with INR > 2.0, thrombocytopenia with platelet counts < 50,000
* Pregnancy (if required a pregnancy test would be performed as part of routine clinical care)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-08; Primary Completion 2017-05-26 (Actual); Study Completion 2017-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Wang, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Focal Cryo Ablation: Subjects with residual barrett's esophagus (less than 3 cm) post ablation will under go one CryoBalloon Focal Ablation treatment
  CryoBalloon Focal Ablation
Period: Overall Study
Arm/Group | Focal Cryo Ablation
Started | 18
Completed | 15
Not Completed | 3
Not completed — Screen Failure | 3

BASELINE CHARACTERISTICS:
Arm/Group | Focal Cryo Ablation
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 67.94 (7.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 16
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 18

OUTCOME MEASURES:

1. Primary Outcome: Eradication of Barrett's Esophagus
Description: Number of subjects to have eradication of barrett's esophagus after Cryoballoon Focal Ablation
Time Frame: 3 months post Cryoballon Focal Ablation
Measure: Count of Participants; unit: Participants
Arm/Group | Focal Cryo Ablation
Number analyzed (Participants) | 15
Participants | 2

ADVERSE EVENTS:
Time Frame: Adverse events were collected from baseline to end of study for a total of approximately 3 months on all participants.
Arm/Group | Focal Cryo Ablation
All-Cause Mortality (participants affected / at risk) | 1/18
Serious Adverse Events (participants affected / at risk) | 0/18
Other Adverse Events (participants affected / at risk) | 1/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Focal Cryo Ablation (N=18)
Difficulty Swallowing (Gastrointestinal disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2016-04-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT02230410/Prot_000.pdf